CLINICAL TRIAL: NCT05600725
Title: Novel Pacing Modality to Initiate Favorable Cardiac Remodeling in Heart Disease
Brief Title: Novel Cardiac Pacing to Initiate Cardiac Remodeling in Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denise Hodgson-Zingman (Other)
Responsible Party: Sponsor-Investigator, Denise Hodgson-Zingman, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202202351
Record Dates: First submitted 2022-06-27; First posted 2022-10-31 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Cardiomyopathies; Heart Rate; Conditioning
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized in a single-blinded fashion to intervention vs. sham treatment
Who Masked: Participant, Outcomes Assessor
Masking Description: Subjects will be unaware of their group assignment. Investigators delivering the intervention vs. sham will be aware. Analysts processing primary data (serum testing, echocardiographic dimensions, 6-min walk distance, CPEX) will not be aware of group assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pacing intervention (Experimental): A novel atrial pacing approach will be delivered using the subject's already implanted pacemaker, ICD or BiV/ICD while the subject is in a semi-recumbent position and while hemodynamic and symptom data is collected. This will be repeated once daily, 3d/wk over 4 weeks.
  Interventions: Other: novel atrial pacing approach
- Sham pacing (Sham Comparator): Subjects in this arm will be treated identically to the subjects in the pacing intervention arm but their already implanted pacemaker, ICD or BiV/ICD will have programming changes simulated but not actually implemented.
  Interventions: Other: sham pacing approach

INTERVENTIONS:
Other: novel atrial pacing approach — See US Patent #10987516. An atrial pacing method that preserves atrioventricular and interventricular synchrony to reproduce an exercise-typical envelope of heart rate.
  Arms: Pacing intervention
Other: sham pacing approach — A pacemaker/ICD interrogator/programmer will be used to simulate changes in pacing rate over the same time period as the intervention group but the programming changes will not actually be implemented and not change in paced heart rate will occur.
  Arms: Sham pacing

SUMMARY:
This project utilizes a novel cardiac pacing approach hypothesized to initiate beneficial cardiac conditioning and remodeling over a period of time.

DETAILED DESCRIPTION:
The project studies subjects with non-ischemic cardiomyopathy who have a pacing device already implanted. Subjects randomized to the pacing intervention versus a sham intervention will be compared for various symptomatic, functional and other outcomes. Each subject will undergo baseline quality of life/symptom questionnaires and clinical testing for cardiac functional/structural effects and exercise tolerance, then the intervention vs. sham (subjects blinded to their category), followed by repeat questionnaires and clinical testing. Medical record review will be undertaken to establish demographic variables, baseline and follow up testing results.

ELIGIBILITY:
Inclusion Criteria:

* Non-Ischemic Cardiomyopathy
* Ejection Fraction </= 35% despite at least 3 months stable standard medical management
* New York Heart Association Class II-III symptoms
* Dual chamber implantable cardioverter defibrillator in place or Biventricular ICD in place (over 3 months old)
* Normal Atrioventricular conduction or Biventricular ICD
* QRS < 120 msec (inherent conduction or paced with BiV ICD)

Exclusion criteria:

* Age < 18 years
* Inability to ambulate safely
* Congenital or primary valve disease
* Left Ventricular thrombus
* Severe peripheral arterial disease
* Admission for life-threatening condition (eg heart failure, stroke) in the past 3 months
* Major surgery in the past 3 months or anticipated during the period of the trial
* Paced or intrinsic QRS >120 msec
* Life expectancy < 1 year
* Hemodialysis
* Hematocrit < 30%
* Severe Chronic lung disease
* Pregnancy
* ICD battery longevity < 1 year
* Unsuppressed atrial arrhythmias
* Already participating in an exercise programusion Criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-11-02 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Quality of life/symptom score | 4 weeks after start of the protocol
  Minnesota Living with Heart Failure Score (range 0-105, higher scores indicate worse quality of life)

SECONDARY OUTCOMES:
systolic blood pressure | every 5 minutes during intervention/sham in weeks 1-4 of the protocol
  systolic blood pressure (mmHg) as a continuous variable
diastolic blood pressure | every 5 minutes during intervention/sham in weeks 1-4 of the protocol
  systolic blood pressure (mmHg) as a continuous variable
Oxygen saturation | every 5 minutes during intervention/sham in weeks 1-4 of the protocol
  oxygen saturation by pulse oximeter (%) as a continuous variable
cardiac output | every 5 minutes during intervention/sham in weeks 1-4 of the protocol
  cardiac output (liters/minute) as measured by thoracic impedance and reported as a continuous variable
MACE | 4 weeks and 4 months after start of the protocol
  Major adverse cardiac events: composite of total death, MI, stroke, hospitalization due to heart failure, revascularization
six minute walk | at the time of enrollment, and at 4 weeks after start of the protocol
  distance ambulated in 6 minutes (meters)

CONTACTS AND LOCATIONS:
Overall Officials: Denice Hodgson-Zingman, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States